CLINICAL TRIAL: NCT00745810
Title: The Effects of Anesthetic Management on Oxidative Injuries After Cardiopulmonary Bypass
Brief Title: Anesthetic Management and Remote Reperfusion Injuries
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200705022R
Record Dates: First submitted 2008-08-31; First posted 2008-09-03 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-06

CONDITIONS: Heart Valve Diseases
Keywords: cardiopulmonary bypass; oxidative injuries
MeSH Terms: conditions — Heart Valve Diseases | interventions — Cardiopulmonary Bypass; Oxidative Stress; Complement System Proteins; Leukocyte Elastase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — whole blood and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: sequential changes before and after cardiopulmonary bypass including ROS, antioxidant status, leukocyte elastase, complements, inflammatory cytokines
  Interventions: Other: Cardiopulmonary bypass

INTERVENTIONS:
Other: Cardiopulmonary bypass — sequential changes of oxidative injuries before and after cardiopulmonary bypass
  Other Names: oxidative injuries; inflammatory cytokines; complements; leukocyte elastase

SUMMARY:
Ischemia- reperfusion ( IR ) injuries were not only seen in the transplanted organs but also the remote organs such as lungs that brings major postoperative complications. Severe complications such as pulmonary infiltration and pulmonary edema following reperfusion were frequently associated with liver transplantation. Cardiac surgery performed with the use of cardiopulmonary bypass ( CPB ) provokes a systemic inflammatory response syndrome that affects postoperative pulmonary, myocardiac and renal functions. Previous study about the reperfusion injuries was focused on the leukocyte and endothelial activation and the following oxidative injuries, however, the alteration on pulmonary function such as dynamic compliance and the oxidative/antioxidative balance in erythrocytes and the following effects in CPB have not been fully studied. Erythrocytes' reaction to oxidative stress including cytoplasma and cell membrane should be studied because RBCs are the major circulating blood cells having different types of antioxidant system to capture reactive oxygen species ( ROS ) thus RBC may be severely injured by ROS or protected ROS injuries during CPB. In these three-year study, we plan to explore the extent and pattern of remote oxidative injuries in lungs by massive ROS production and the following products released from reperfused organs. In the first year, the remote pulmonary injuries from hepatic IR will be focused. We plan to establish an animal model for pulmonary function and pulmonary injury assessments including dynamic compliance (Cdyn), pulmonary edema wet-to-dry ratio (W/D), malondialdehyde (MDA) and histopathological findings under hepatic IR challenge. In the second year, the IR effects during and after CPB on circulating blood cells will be fully studied. We plan to investigate the magnitude, subtypes and timing on ROS production, the changes of oxidative and antioxidant activities of erythrocytes including cytoplasma and cell membrane, the changes on leukocytes and plasma to explore the roles of circulating erythrocytes on oxidative stress in CPB. In the third year, we plan to try propofol, stated having antioxidant in vivo and in vitro, on the remote pulmonary injuries following hepatic IR and CPB.

DETAILED DESCRIPTION:
Seven ml blood sample were taken from arterial line after stabilization of anesthesia (T1), 30 minutes after total CPB (T2), one hour after weaning from CPB (T3) and 24 hours after weaning from CPB (T4). One ml blood sample was immediately wrapped in aluminum foil and kept in ice to immediate measurements of MetHb, COHb and CL (ROS). CL assay was carried out within 2 hours of sampling. Six ml samples remained was placed into tubes containing ethylenediamine tetraacetic acid. Serum were separated ( at 2000rpm for 10 minutes) immediately after sampling and stored at -80℃ for TAS assay, cytokine measurements, malondialdehyde (MDA) determination, complements and leukocyte elastase measurements. Those assay and measurements were carried out within 4 weeks of surgery.

Measurements of hemoglobin (Hb), COHb and MetHb: Hb, COHb and MetHb were measured immediately with ABL520, Radiometer, Copenhagen, Denmark).

Measurement of Redox balance: 0.2ml of fresh drawn blood was used to measure ROS production by lucigenin Chemiluminescence (CL) (detecting superoxide mainly) and luminal CL (detecting H2O2 and HOCl mainly) as previous study.The total antioxidant status in 20 uL of plasma was measured with a total antioxidant status (TAS) kit ( TAS CAL, Randox). Hemodilution effects with CPB, TAS levels at T2 were corrected with the hematocrits. Lipid peroxidation was determined by the thiobarbiturate reaction measuring the formation of MDA in plasma by TBARS assay kit (Cayman chemical co. USA) Cytokines analysis: Inflammatory cytokines were analysis with RayBio human inflammation antibody array 3 according to the manufacturer's instruction. (Cat# AAH-INF-3, RayBiotech Inc. Norcross, GA, USA).29 Measurements of complement activation and leukocytes activation: Complement Component 3a (C3a), C5a, and Human Terminal Complement Complex C5b-9 (C5b-9) were measured with human C3a EIA kit, human C5a EIA kit, Human Terminal Complement Complex C5b-9 kit, Life Science Inc.). Leukocyte elastase were measured by Elisa kit for Human Elastase 2,Neutrophil(NE, Life Science Inc.)

ELIGIBILITY:
Inclusion Criteria:

* age > 20 y/0, need cardiopulmonary bypass

Exclusion Criteria:

* severe anemia, hematologic diseases, hormone therapy, previous valvular surgery, blood transfusion in recent 3 months

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who receive an open heart surgery under cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ya-jung cheng, PhD, Principal Investigator — Department of anesthesia, national taiwan university hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan